CLINICAL TRIAL: NCT01352702
Title: Impact of Dabigatran and Phenprocoumon on Clopidogrel Mediated ADP Induced Platelet Aggregation in Patients With Atrial Fibrillation
Acronym: Dabi-ADP-2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment; Study was terminated for futility reasons
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. A01711; 2011-000504-18 (EudraCT Number)
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Heart Disease; Atrial Fibrillation; Acute Coronary Syndrome; Atherosclerosis
MeSH Terms: conditions — Coronary Disease; Atrial Fibrillation; Acute Coronary Syndrome; Atherosclerosis | interventions — Dabigatran; Phenprocoumon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Dabigatran Therapy
  Interventions: Drug: Dabigatran
- Arm 2 (Active Comparator): Phenprocoumon Therapy
  Interventions: Drug: Phenprocoumon

INTERVENTIONS:
Drug: Dabigatran — Patients assigned to this group will receive Dabigatran
  Other Names: Pradaxa
  Arms: Arm 1
Drug: Phenprocoumon — Patients assigned to this group will receive Phenprocoumon
  Other Names: Marcumar
  Arms: Arm 2

SUMMARY:
The aim of this study is to evaluate whether dabigatran reduces clopidogrel mediated ADP induced platelet aggregation measured by MEA as compared to phenprocoumon after a two-week treatment with either agent.

DETAILED DESCRIPTION:
Oral anticoagulation with vitamin K antagonists (OAC) is the standard care for reducing stroke in patients with atrial fibrillation. Just recently the direct, competitive thrombin inhibitor dabigatran has been approved by the FDA for stroke prevention in patients with atrial fibrillation. In a large multicenter trial it was shown that dabigatran was at least as effective as Vitamin K antagonists in the prevention of stroke without an increase of major hemorrhage.

Approximately 6 % of patients who undergo coronary stenting and need DAT with aspirin and clopidogrel need in addition OAC for the reduction of cardiac, cerebral and systemic thromboembolic events5. These patients will therefore need triple therapy, a therapy which is associated with increased bleeding complications. Although phenprocoumon given solely without clopidogrel has no impact on ADP induced platelet aggregation, it has been shown that phenprocoumon significantly attenuates the antiplatelet effects of clopidogrel.

ADP induced platelet aggregation measured with multiple electrode platelet aggregometry (MEA) is a marker for the efficacy of the clopidogrel therapy and (i) a low response (AUC ≥ 468) to clopidogrel has been associated with an increase of ischemic events such as stent thrombosis and (ii) patients with an enhanced response to clopidogrel (AUC ≤ 188) have higher bleeding rates.

It is therefore crucial to evaluate whether an additional antithrombotic therapy such as dabigatran alters clopidogrel mediated ADP induced platelet aggregation. While it has been shown that intravenous administration of the direct thrombin inhibitor bivalirudin further reduces ADP induced platelet aggregation in patients on clopidogrel therapy, it is unknown whether dabigatran has also an impact on ADP induced platelet aggregation.

To evaluate the impact of dabigatran on ADP induced platelet aggregation we will randomize patients with atrial fibrillation and the need for oral anticoagulation and current clopidogrel therapy for a two-week treatment with either dabigatran or phenprocoumon and we hypothesize that dabigatran is superior to phenprocoumon in the reduction of ADP induced platelet aggregation. Patients who are not concomitantly treated with clopidogrel are being studied in a different trial with a similar study design (Dabi ADP-1).

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with atrial fibrillation and an indication for oral anticoagulation (CHA2DS2-VASc score≥ 1).
* Current clopidogrel treatment
* Informed, written consent by the patient or her/his legally-authorized representative for participation in the study.

Key Exclusion Criteria:

* Age ≤18 years
* Cardiogenic shock
* Current therapy with dabigatran
* Patients with a recent thromboembolic event and high thromboembolic risk requiring bridging therapy with either unfractionated heparin or LMWH
* Contraindication for oral anticoagulation
* Active bleeding
* Known allergy or intolerance to the study medications: dabigatran, phenprocoumon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
ADP induced platelet aggregation | 2 weeks
  To determine whether there are differences in ADP induced platelet aggregation after 2 weeks in patients receiving dabigatran or phenprocoumon.

SECONDARY OUTCOMES:
Platelet function tests | 2 weeks
  ADPtest HS (MEA) , TRAP, Collagen
Coagulation parameters | 2 weeks
  aPTT, INR, Thrombin coagulation time

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Principal Investigator — Deutsches Herzzentrum München, Klinik für Herz- und Kreislauferkrankungen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany